CLINICAL TRIAL: NCT02111707
Title: Timing of Indomethacin Administration for the Prevention of Post-ERCP Pancreatitis (PEP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00041158
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin

ARMS (2):
- Rectal Indomethacin pre-ERCP (Active Comparator): Patients will receive rectal indomethacin 100mg 30 minutes before procedure (ERCP).
  Interventions: Drug: Rectal indomethacin 100mg one time before or after ERCP
- Rectal Indomethacin post-ERCP (Active Comparator): Patients will receive rectal indomethacin 100mg immediately after procedure (ERCP)
  Interventions: Drug: Rectal indomethacin 100mg one time before or after ERCP

INTERVENTIONS:
Drug: Rectal indomethacin 100mg one time before or after ERCP — Patients will receive rectal indomethacin suppository 30 minutes before or immediately after ERCP for prevention of post-procedure pancreatitis. Patients will be randomized to the timing of administration.
  Other Names: Indocid 100mg

SUMMARY:
To determine if the timing of administration of indomethacin affects the primary outcome of post-ERCP pancreatitis (PEP). Patients undergoing ERCP will be randomly assigned to receive pre or post-procedure rectal indomethacin to prevent the occurrence of PEP.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for ERCP at the University of Alberta
* Age greater than 18 years
* Ability to provide written informed consent

Exclusion Criteria:

* Acute pancreatitis
* Active peptic ulcer disease
* Rectal disease
* Aspirin-induced asthma
* Nonsteroidal anti-inflammatory drug (NSAIDs) induced hypersensitivity
* Pregnancy
* Breast feeding
* Creatinine clearance < 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Rate of Post-ERCP pancreatitis | 30 days

SECONDARY OUTCOMES:
Severity of Post-ERCP pancreatitis | 30 days
  To evaluate the severity of post-ERCP pancreatitis between the 2 groups studied

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Sotoudehmanesh R, Khatibian M, Kolahdoozan S, Ainechi S, Malboosbaf R, Nouraie M. Indomethacin may reduce the incidence and severity of acute pancreatitis after ERCP. Am J Gastroenterol. 2007 May;102(5):978-83. doi: 10.1111/j.1572-0241.2007.01165.x. Epub 2007 Mar 13. PMID 17355281
- [Result] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Result] Murray B, Carter R, Imrie C, Evans S, O'Suilleabhain C. Diclofenac reduces the incidence of acute pancreatitis after endoscopic retrograde cholangiopancreatography. Gastroenterology. 2003 Jun;124(7):1786-91. doi: 10.1016/s0016-5085(03)00384-6. PMID 12806612
- [Result] Montano Loza A, Rodriguez Lomeli X, Garcia Correa JE, Davalos Cobian C, Cervantes Guevara G, Medrano Munoz F, Fuentes Orozco C, Gonzalez Ojeda A. [Effect of the administration of rectal indomethacin on amylase serum levels after endoscopic retrograde cholangiopancreatography, and its impact on the development of secondary pancreatitis episodes]. Rev Esp Enferm Dig. 2007 Jun;99(6):330-6. doi: 10.4321/s1130-01082007000600005. Spanish. PMID 17883296